CLINICAL TRIAL: NCT03522493
Title: The Effect of Age and Inspiratory Resistance on the Inspiratory Gas Levels While Wearing Air Purifying Respirator "Yaalom Katom"
Brief Title: The Effect of Age and Inspiratory Resistance on the Inspiratory Gas Levels While Wearing Air Purifying Respirator "
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical Corps, Israel Defense Force (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1552-2015
Record Dates: First submitted 2016-04-07; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Aging

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Young group (Active Comparator): This arm include 20 young subjects that will perform the same experiment as the old group for a comparison reasons.
  Interventions: Device: "Yaalom Katom"
- Old group (Experimental): This group us the group of interest. This group will wear the mask and is expected to show differences from the younger group.
  Interventions: Device: "Yaalom Katom"

INTERVENTIONS:
Device: "Yaalom Katom" — Full face Gas mask

SUMMARY:
20 healthy young subjects and 20 healthy older subjects will go through a medical examination. Subjects will be asked for their medical history especially on respiratory and cardiac diseases. All subjects will go through a spirometry test to evaluate their respiratory function. After their medical clearance each subjects will be asked to wear a CBRN respirator for 45 minutes. 15 minutes without filter, 15 minute with 0.8 cmH2O resistance, and 15 minutes with 1.2 cmH2O resistance. Throughout the test, Pco2 AND PO2 will be measured. The investigator will evaluate the effect of resistance (filter resistance) and the age of the subject on CO2 accumulation in the mask.

DETAILED DESCRIPTION:
After signing the consent form, 20 healthy young subjects and 20 healthy older subjects will go through a medical examination. Subjects will be asked for their medical history especially on respiratory and cardiac diseases. All subjects will go through a spirometry test to evaluate their respiratory function. After their medical clearance each subjects will be asked to wear a CBRN respirator for 45 minutes. 15 minutes without filter, 15 minute with 0.8 cmH2O resistance, and 15 minutes with 1.2 cmH2O resistance. Throughout the test, Pco2 AND PO2 will be measured with mass spectrometer. Oxygen saturation, Pulse rate, and minute ventilation will also be monitored. The investigator will evaluate the effect of resistance (filter resistance) and the age of the subject on CO2 accumulation in the mask.

ELIGIBILITY:
Inclusion Criteria:

Healthy females and males, with no respiratory, cardio vascular diseases, high blood pressure, psychiatric problem, degenerative nervous system problem, and chronic head ache, muscular disease, or severe acute disease within the two weeks before the study. age 18 and 25, and 55 and 70 years old. Who volunteer to the study

-

Exclusion Criteria:

Did not pass the Inclusion criteria, pregnant women, O2 saturation lower then 95%, pathological sound from the heart or lungs. Claustrophobia, smoking history more then 2.5 packs years.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Average CO2 (%) | 45 minutes
  Average CO2 (%) will be measured continusly during each of the filters for the two groups.

SECONDARY OUTCOMES:
Respiratory discomfort (borg scale 1-10) | 45 minutes
  Respiratory discomfort will be measured using the Borg scale for each filters and for the two groups
Average O2 (%) | 45 minutes
  Average O2 (%) will be measured continusly during each of the filters for the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Israel Naval Medical Institute, Haifa, Israel